CLINICAL TRIAL: NCT01076075
Title: A Phase III, Randomized, Clinical Trial to Evaluate the Safety and Efficacy of the Addition of Sitagliptin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on a Sulfonylurea in Combination With Metformin
Brief Title: A Study to Evaluate the Safety and Efficacy of Sitagliptin 100 mg in Participants With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control (MK-0431-229)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-229; 2010_513; MK-0431-229 (Other: protocol number)
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Pioglitazone; glimepiride; Gliclazide; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo/pioglitazone (Active Comparator): Phase A (Weeks 0-24): placebo to Sitagliptin 100 mg; Phase B (Weeks 24-54): placebo to Sitagliptin 100 mg + pioglitazone 30 mg
  Interventions: Drug: Comparator: placebo to Sitagliptin; Drug: Comparator: pioglitazone; Drug: Glimepiride or gliclazide; Drug: Metformin; Drug: Pioglitazone rescue therapy
- Sitagliptin (Experimental): Phase A (Weeks 0-24): Sitagliptin 100 mg; Phase B (Weeks 24-54): Sitagliptin 100 mg + placebo to pioglitazone
  Interventions: Drug: Sitagliptin phosphate; Drug: Comparator: placebo to pioglitazone; Drug: Glimepiride or gliclazide; Drug: Metformin; Drug: Pioglitazone rescue therapy

INTERVENTIONS:
Drug: Sitagliptin phosphate — Phase A (Weeks 0-24): Sitagliptin 100 mg once a day for 24 weeks; Phase B (Weeks 24-54): Sitagliptin 100 mg once a day for 30 weeks
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Comparator: placebo to pioglitazone — Phase B (Weeks 24-54): placebo to pioglitazone 30 mg once a day for 30 weeks
  Arms: Sitagliptin
Drug: Comparator: placebo to Sitagliptin — Phase A (Weeks 0-24): placebo to Sitagliptin 100 mg once a day for 24 weeks; Phase B (Weeks 24-54): placebo to Sitagliptin once a day for 30 weeks
  Arms: placebo/pioglitazone
Drug: Comparator: pioglitazone — Phase B (Weeks 24-54): pioglitazone 30 mg once a day for 30 weeks
  Other Names: Actos;
  Arms: placebo/pioglitazone
Drug: Glimepiride or gliclazide — Phase A (Weeks 0-24): stable dose, as prescribed by investigator, of glimepiride or gliclazide; Phase B (Weeks 24-54): stable dose, as prescribed by investigator, of glimepiride or gliclazide
Drug: Metformin — Phase A (Weeks 0-24): stable dose, as prescribed
  by investigator, of metformin; Phase B (Weeks 24-
  54): stable dose, as prescribed by investigator, of
  metformin
Drug: Pioglitazone rescue therapy — Phase A (Weeks 0-24): participants not meeting specific glycemic goals will receive pioglitazone (open label) at a dose determined by the investigator. These participants will not initiate Phase B (Weeks 24-54) double blind pioglitazone.
  Other Names: Actos

SUMMARY:
This study will evaluate whether the addition of Sitagliptin treatment provides a greater decrease in A1C levels compared to placebo in participants with inadequate glycemic control on sulfonylurea and metformin combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Hemoglobin A1C of ≥7.5% and ≤10.5%
* Currently taking a stable dose of metformin (at least 1500 mg/day) and either glimepiride (at least 2 mg/day) or gliclazide (at least 50% of maximum registered dose) for at least 10 weeks prior to study start
* Male, or a female who is highly unlikely to conceive

Exclusion Criteria:

* Type 1 diabetes mellitus or ketoacidosis
* Taking a dipeptidyl peptidase-4 (DPP-4) inhibitor (such as sitagliptin) or a glucagon-like peptide-1 (GLP-1) mimetic (such as exenatide or liraglutide) or required insulin therapy within 12 weeks prior to study start
* On a weight loss program not in the maintenance phase or on a weight loss medication
* History of liver disease, heart failure, heart disease, stroke, high blood pressure, blood disorders, or cancer
* HIV positive
* Pregnant

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2010-06-03 (Actual); Primary Completion 2011-07-11 (Actual); Study Completion 2012-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Moses RG, Round E, Shentu Y, Golm GT, O'neill EA, Gantz I, Engel SS, Kaufman KD, Goldstein BJ. A randomized clinical trial evaluating the safety and efficacy of sitagliptin added to the combination of sulfonylurea and metformin in patients with type 2 diabetes mellitus and inadequate glycemic control. J Diabetes. 2016 Sep;8(5):701-11. doi: 10.1111/1753-0407.12351. Epub 2016 Feb 3. PMID 26625270

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 762 participants were screened, 335 participants were excluded, and 427 participants were randomized. There was a single-blind run-in prior to randomization.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo/Pioglitazone
Started | 213 (3 participants were excluded from safety and efficacy analyses due to one site's non-compliance) | 214 (2 participants were excluded from safety and efficacy analyses due to one site's non-compliance)
Completed Phase A | 199 | 189
Completed | 172 | 167
Not Completed | 41 | 47
Not completed — Adverse Event | 3 | 9
Not completed — Lack of Efficacy | 5 | 4
Not completed — Lost to Follow-up | 6 | 5
Not completed — other | 19 | 9
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 8 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo/Pioglitazone | Total
Number analyzed (Participants) | 210 | 212 | 422
Age, Continuous [Mean (Standard Deviation); unit: years] — Number of Baseline Participants for Sitagliptin (210) and for Placebo/Pioglitazone (212). Five participants (Sitagliptin: 3, Placebo/Pioglitazone: 2) were excluded from analyses due to one site's non-compliance.
  years | 54.4 (9.6) | 55.4 (10.2) | 54.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of Baseline Participants for Sitagliptin (210) and for Placebo/Pioglitazone (212). Five participants (Sitagliptin: 3, Placebo/Pioglitazone: 2) were excluded from analyses due to one site's non-compliance.
  Participants
    Female | 115 | 114 | 229
    Male | 95 | 98 | 193
Hemoglobin A1C [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] — Number of Baseline Participants for Sitagliptin (210) and for Placebo/Pioglitazone (212). Five participants (Sitagliptin: 3, Placebo/Pioglitazone: 2) were excluded from analyses due to one site's non-compliance.
  Percentage of glycosylated hemoglobin | 8.4 (0.8) | 8.4 (0.9) | 8.4 (0.8)
2-Hour Post-Meal Glucose [Mean (Standard Deviation); unit: mg/dL] — Number of Baseline Participants for Sitagliptin (202) and for Placebo/Pioglitazone (208). Five participants (Sitagliptin: 3, Placebo/Pioglitazone: 2) were excluded from analyses due to one site's non-compliance.
  mg/dL | 240.3 (60.6) | 243.3 (68.8) | 241.8 (64.8)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — Number of Baseline Participants for Sitagliptin (210) and for Placebo/Pioglitazone (212). Five participants (Sitagliptin: 3, Placebo/Pioglitazone: 2) were excluded from analyses due to one site's non-compliance.
  mg/dL | 164.8 (40.8) | 165.0 (43.9) | 164.9 (42.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (%) at Week 24
Description: Change from baseline reflects the Week 24 value minus the baseline value. A1C represents the percentage of glycosylated hemoglobin.
Time Frame: Baseline and Week 24
Population: The Full Analysis Set Population received at least one dose of study treatment and had baseline data and at least one post-baseline treatment endpoint observation for the analysis endpoint. Missing data were imputed using last observation carried forward (LOCF). Five participants were excluded from analyses due to one site's non-compliance.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of glycosylated hemoglobin
Groups:
- Sitagliptin: Phase A (Weeks 0-24): Sitagliptin 100 mg
- Placebo/Pioglitazone: Phase A (Week 0-24): Placebo to Sitagliptin 100 mg
Arm/Group | Sitagliptin | Placebo/Pioglitazone
Number analyzed (Participants) | 203 | 202
Percentage of glycosylated hemoglobin | -0.84 (0.82) [-0.97 to -0.71] | -0.16 (0.84) [-0.28 to -0.03]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo/Pioglitazone; Pairwise comparison - Sitagliptin vs. Placebo, using the difference in the Least Squares Means; Test type: Superiority or Other; p < 0.001, ANCOVA; Based on an ANCOVA model controlling for treatment, stratum (type of sulfonylurea) and baseline value; Difference in Least Squares Means = -0.68, 95% CI 2-sided [-0.87 to -0.50]

2. Secondary Outcome: Change From Baseline in 2-hour Post-Meal Glucose at Week 24
Description: Change from baseline reflects the Week 24 value minus the baseline value. Two-hour post-meal glucose was measured following a standard meal.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Sitagliptin: Phase A (Week 0-24): Sitagliptin 100 mg
Arm/Group | Sitagliptin | Placebo/Pioglitazone
Number analyzed (Participants) | 184 | 183
mg/dL | -36.8 (60.8) [-45.2 to -28.4] | -3.3 (67.8) [-11.7 to 5.0]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo/Pioglitazone; Pairwise comparison - Sitagliptin vs. Placebo, difference in the Least Squares Means; Test type: Superiority or Other; p < 0.001, ANCOVA; Based on an ANCOVA model controlling for treatment, stratum (type of sulfonylurea) and baseline value; Difference in Least Squares Means = -33.5, 95% CI 2-sided [-45.3 to -21.7]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 24
Description: Change from baseline reflects the Week 24 value minus the baseline value.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo/Pioglitazone
Number analyzed (Participants) | 204 | 203
mg/dL | -13.2 [-18.8 to -7.7] | 5.3 [-0.2 to 10.9]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo/Pioglitazone; Pairwise comparison - Sitagliptin vs. Placebo, using the difference in the Least Squares Means; Test type: Superiority or Other; p < 0.001, ANCOVA; Based on an ANCOVA model controlling for treatment, stratum (type of sulfonylurea) and baseline value; Difference in Least Squares Means = -18.6, 95% CI 2-sided [-26.4 to -10.7]

4. Primary Outcome: Number of Participants With One or More Adverse Events (AEs) - Week 0 to Week 54
Time Frame: Week 0 to Week 54
Population: The All Patients as Treated Population took at least one dose of study drug. Participants received glycemic rescue medication if they met specific glycemic goals up to Week 24. Adverse events include those that occurred prior to a receiving rescue medication. Five participants were excluded from analyses due to 1 site's non-compliance.
Measure: Number; unit: participants
Groups:
- Placebo/Pioglitazone: Phase A (Weeks 0-24: Placebo to Sitagliptin 100 mg; Phase B (Weeks 24-54): Placebo to Sitagliptin 100 mg + Pioglitazone 30 mg
Arm/Group | Sitagliptin | Placebo/Pioglitazone
Number analyzed (Participants) | 210 | 212
participants | 120 | 122

5. Primary Outcome: Number of Participants Discontinuing Study Drug Due to An Adverse Event
Time Frame: Week 0 to Week 54
Population: The All Patients as Treated Population took at least 1 dose of study drug. Participants received glycemic rescue medication if they met specific glycemic goals up to Week 24. Participants discontinued due to adverse events are reported regardless of rescue medication. Five participants were excluded from analyses due to 1 site's non-compliance.
Measure: Number; unit: participants
Arm/Group | Sitagliptin | Placebo/Pioglitazone
Number analyzed (Participants) | 210 | 212
participants | 3 | 9

ADVERSE EVENTS:
Time Frame: Week 0 to Week 54
Description: All Patients as Treated Population took at least 1 dose of study drug. Participants received glycemic rescue medication if they met specific glycemic goals up to Week 24. Serious AEs (SAEs) are reported regardless of rescue medication. Other AEs are those that occurred prior to rescue medication. Five participants were excluded from analyses.
Arm/Group | Sitagliptin | Placebo/Pioglitazone
Serious Adverse Events (participants affected / at risk) | 6/210 | 9/212
Other Adverse Events (participants affected / at risk) | 49/210 | 44/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=210) | Placebo/Pioglitazone (N=212)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=210) | Placebo/Pioglitazone (N=212)
Upper respiratory tract infection (Infections and infestations) | 14 (15) | 15 (16)
Hypoglcaemia (Metabolism and nutrition disorders) | 38 (187) | 31 (148)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.